CLINICAL TRIAL: NCT06122909
Title: The Effect Of Resuscitation Guided By Two Different Dynamic Parameters On Time To Normalization Of The Capillary Refill Time In Adult Patients With Septic Shock, A Randomized Controlled Prospective Study
Brief Title: The Effect Of Resuscitation Guided By Two Different Dynamic Parameters On Time To Normalization Of The Capillary Refill Time In Adult Patients With Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD ∕ 22.06.664
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Resuscitation
Keywords: capillary refill time; septic shock; resuscitation; ultrasound; dynamic
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Left ventricular outflow tract-velocity time integral (LVOT-VTI) resuscitation based group Inferior vena cava (IVC) diameter variation resuscitation based group
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blinded to the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VTI (Experimental): Group VTI (n=45): will receive resuscitation guided by LVOT-VTI variation after PLR test.
  Interventions: Drug: Group VTI
- Group IVC (Active Comparator): Group IVC (n=45): will receive resuscitation guided by IVC diameter variation after PLR test.
  Interventions: Drug: Group IVC

INTERVENTIONS:
Drug: Group VTI — Group VTI will receive resuscitation guided by LVOT-VTI variation after PLR test.
  Arms: Group VTI
Drug: Group IVC — Group IVC will receive resuscitation guided by IVC diameter variation after PLR test.
  Arms: Group IVC

SUMMARY:
The aim of this study is to compare the effect of resuscitation guided by Left ventricular outflow tract-velocity time integral (LVOT-VTI) variation versus the effect of resuscitation guided by inferior vena cava (IVC) variation on time to normalization of the capillary refill time in adult patients with septic shock, amount of resuscitation fluids, rate of vasopressor and ICU length of stay.

DETAILED DESCRIPTION:
Capillary refill time will be measured by applying firm pressure to the ventral surface of the right index finger distal phalanx with a glass microscope slide. The pressure will be increased until the skin is blank and then maintained for 10 seconds. The time for return of the normal skin color will be registered with a chronometer. A CRT > 3 seconds will be considered abnormal.

Patients with normal CRT at baseline will proceed to periodic monitoring (every hour/6 hours) and start the algorithm if CRT becomes abnormal at any of these timepoints. Patients with abnormal CRT will follow the loop when fulfilling the Sepsis-3 definition of septic shock.

Sepsis time 0 is defined as the time of admission to the ICU for sepsis treatment upon the inclusion criteria. For patients already in the ICU, sepsis time 0 is considered the earliest time at which the patients satisfy the inclusion criteria.

Fluid responsiveness FR will be assessed using a structured approach. Dynamic predictors of FR will be evaluated depending on the individual status, i.e., considering if under MV or spontaneous breathing, Vt, respiratory rate (RR), respiratory system compliance and the presence of arrhythmias.

Passive leg raise PLR is performed by tilting a patient from a 45-degree semi-recumbent head-up position to a 30-45° degree leg-up position or by lifting the legs passively from the horizontal position. This maneuver transfers up to 300 mL of blood from the lower limbs and the splanchnic territory into the intrathoracic compartment and induces significant changes in cardiac preload, mean systemic pressure and the upstream pressure of systemic venous return. It is reliable and can be implemented in either spontaneously breathing or mechanically ventilated patients and can often be repeated. A method that has been recommended by the Surviving Sepsis Campaign, and is appraised by the European Society of Intensive Care Medicine.

After informed consent is obtained from the caregiver, transthoracic two-dimensional 2D, M-mode, and Doppler echocardiography will be performed on commercially available echocardiographic equipment (Mindray, M7 Premium) using a (SP5-1s) probe. Echocardiography will be performed to measure the LVOT diameter measured in the long-axis parasternal view, and the time-velocity integral of the flow wave across the aortic valve (VTI) will be obtained by pulsed wave Doppler and averaged over the whole respiratory cycle. Synchronization of the measurements with the different times of the ventilatory cycle will be verified by insertion of a pressure signal.

For the spontaneously breathing patients, the images will be obtained over 1 respiratory cycle, inspiration and expiration will be defined by the biggest and smallest size, respectively. Multiple ECHO images will be obtained and the 3 most consistent will be averaged off-line.

LVOT-VTI variation and IVC diameter variation will be measured twice at least for every patient in both groups at baseline and post PLR. The 3 most consistent recordings will be chosen and averaged at baseline and post PLR for the sake of precision of values.

IVC Collapsibility diameter < 21 mm and index ≥ 50% indicates fluid responsiveness in spontaneously breathing patients. IVC distensibility index > 18% indicates fluid responsiveness in mechanically ventilated patients. Passive leg raising test > 12% increase in SV indicates fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* adult patients ( ≥ 18 years) of either gender with septic shock according to the Sepsis-3

Exclusion Criteria:

* Known history of any cardiac pathology, acute coronary syndrome, cardiac dysrhythmias (as a primary diagnosis), acute pulmonary edema or known poor systolic cardiac function (left ventricular ejection fraction < 50%).
* Body mass index ≥ 35 kg/m2 .
* Concomitant acute respiratory distress syndrome) or high PEEP (> 10 cmH2O) requirements on mechanical ventilation (MV).
* Child B or C liver cirrhosis.
* End-stage renal disease with or without dialysis.
* Pregnancy.
* Multi-organ system failure.
* Active hemorrhage.
* Head trauma.
* Intra-abdominal hypertension (> 15 mmHg).
* Declined to consent.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Time to normalization of the capillary refill time (≤ 3 sec) | 12 hours
  Time to normalization of the capillary refill time (≤ 3 sec.) in adult patients with septic shock at 6h of septic shock recognition in patients with delayed capillary refill time (> 3 sec.)

SECONDARY OUTCOMES:
Amount of resuscitation fluids | 24 hours
  total amount of lactated ringer crystalloid solution resuscitation
Total amount of vasopressors. | 24 hours
  Total amount of vasopressors.
Change in Creatinine-based Kidney Disease: Improving Global Outcome (KDIGO) score | 72 hours
  Change in Creatinine-based Kidney Disease: Improving Global Outcome (KDIGO) score from baseline KDIGO score:Stage 1 Serum creatinine 1.5-1.9 times baseline or ≥0.3 mg/dl (≥26.5 mmol/l) increase or Urine output <0.5 ml/kg/h for 6-12 hours
  Stage 2 Serum creatinine 2.0-2.9 times baseline or <0.5 ml/kg/h for ≥12 hours
  Stage 3 Serum creatinine 3.0 times baseline or Increase in serum creatinine to ≥4.0 mg/dl (≥353.6 mmol/l) or Initiation of renal replacement therapy or in patients <18 years, decrease in eGFR to <35 ml/min per 1.73 m² or Urine output <0.3 ml/kg/h for ≥24 hours or anuria for ≥12 hours
ICU length of stay | 1 week
  ICU length of stay from admission to discharge from ICU.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura University, Central Hospital, Al Mansurah, Dakahlia Governorate
  - Cairo university hospitals, kasralainy, Cairo

IPD SHARING:
Plan to Share IPD: No